CLINICAL TRIAL: NCT03913195
Title: A Phase 3 Study of the Safety of Trogarzo® Administered as an Undiluted "IV Push" Over a Reduced Interval or as an Intramuscular Injection in Clinically Stable HIV-1 Infected Trogarzo® Experienced Patients and Healthy HIV-uninfected Volunteers
Brief Title: Study of the Safety of Trogarzo™ Administered as an Undiluted "IV Push" or an Intramuscular Injection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TaiMed Biologics Inc. (Industry)
Collaborators: Westat (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TMB-302
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: HIV-1-infection
Keywords: HIV; ibalizumab; Multi-drug Resistant (MDR) HIV
MeSH Terms: interventions — ibalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Sentinel Group-HIV + (Experimental): Five (5) participants will receive two successive doses of 800mg ibalizumab administered in accordance with the prescribing information followed by five (5) successive 800mg doses on a schedule gradually increasing drug concentration and decreasing administration time.
  Interventions: Drug: ibalizumab-uiyk
- Core Group- HIV+ (Experimental): HIV-infected Core Group participants will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via undiluted IV Push over 30 seconds.
  Interventions: Drug: ibalizumab-uiyk
- Core Group-HIV uninfected (Experimental): Healthy Volunteer Core Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via undiluted IV Push over 30 seconds.
  Interventions: Drug: ibalizumab-uiyk
- Intramuscular Injection Group-HIV+ (Experimental): HIV+ participants in this group will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via intramuscular injection.
  Interventions: Drug: ibalizumab-uiyk
- Intramuscular Injection Group-HIV uninfected (Experimental): Healthy Volunteer Intramuscular Injection Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via intramuscular injection.
  Interventions: Drug: ibalizumab-uiyk

INTERVENTIONS:
Drug: ibalizumab-uiyk — Ibalizumab-uiyk is an Immunoglobulin G4 (IgG4) monoclonal antibody targeting domain 2 of the extracellular portion of the Cluster of Differentiation 4 (CD4) protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
  Other Names: Trogarzo

SUMMARY:
This study is designed to assess the safety and pharmacokinetic profile of 800 mg Trogarzo once every two weeks administered via "IV Push" or intramuscular injection. An initial "Sentinel Group" of 5 participants will begin receiving 800mg Trogarzo on a gradual schedule of increasing concentration and decreasing administration time until undiluted IV Push over 30 seconds is achieved, while safety and pharmacokinetics are evaluated. If no safety signals are seen, the Core Group of 15 participants will be enrolled. The Core Group will receive 800mg Trogarzo via undiluted IV Push over 30 seconds while safety and pharmacokinetics are monitored. After completion of the IV Push portion of the study, a second group of 20 participants will be enrolled to evaluate the safety and pharmacokinetics of administration of 800mg via intramuscular injection.

DETAILED DESCRIPTION:
This goal of this Phase 3 is to evaluate the safety and pharmacokinetics of administering Trogarzo 800 mg once every two weeks as an undiluted IV Push over 30 seconds, and as an intramuscular injection in clinically stable HIV-1 infected patients currently receiving treatment with a stable Trogarzo-containing regimen and in healthy volunteers.

The first five (5) patients enrolled will comprise the Sentinel Group. Patients six (6) through twenty (20) (the Core Group) will not be screened until the Sentinel Group has completed Day 99 (14 weeks) of the study and the DSMB has reviewed the data accumulated and given approval for enrollment of the Core Group to proceed.

The Sentinel Group will receive 2 successive doses of Trogarzo in accordance with the prescribing information. Safety and pharmacokinetic data from these administrations will serve as the comparator for each study participant. Beginning at Day 29 and continuing through Day 85, Sentinel Group participants will begin receiving the prescribed dosage of Trogarzo once every two weeks through Day 85 of the study on a schedule of increasing drug concentration and decreasing administration time at each visit to achieve an undiluted IV Push administration of Trogarzo over 30 seconds.

After review of data from the Sentinel Group by a Data Safety Monitoring Board (DSMB), if approved the study will continue with enrollment of the Core Group, which will enroll both clinically stable HIV-infected patients on a stable Trogarzo-containing treatment regimen and healthy volunteers. The HIV-infected participants in the Core Group will receive 2 successive doses of Trogarzo in accordance with the prescribing information. Safety and pharmacokinetic data from these administrations will serve as the comparator for each study participant. Thereafter, HIV-infected participants in the Core Group will receive the prescribed dosage of Trogarzo via undiluted IV Push over 30 seconds through Day 71 of the study.

Healthy Volunteers in the Core Group will receive a single loading dose of 2000mg of Trogarzo, followed by three successive doses of 800mg Trogarzo in accordance with the prescribing information in order to reach steady state before pharmacokinetic data for analysis are collected. Thereafter, Healthy Volunteers in the Core Group will follow the same schedule of drug administration and assessments as the HIV-infected participants in the Core Group.

HIV-infected participants in the Intramuscular Injection Group will receive 2 successive doses of Trogarzo in accordance with the prescribing information. Safety and pharmacokinetic data from these administrations will serve as the comparator for each study participant. Thereafter, HIV-infected Intramuscular Injection Group participants will receive the prescribed dosage of Trogarzo via intramuscular injection beginning at Day 29 and continuing through Day 71.

Healthy Volunteers in the Intramuscular Injection Group will receive a single loading dose of 2000mg of Trogarzo, followed by three successive doses of 800mg Trogarzo in accordance with the prescribing information in order to reach steady state before pharmacokinetic data for analysis are collected. Thereafter, Healthy Volunteers in the Intramuscular Injection Group will follow the same schedule of drug administration and assessments as the HIV-infected participants in the Intramuscular Injection Group.

ELIGIBILITY:
Inclusion Criteria - HIV-infected participants (all groups):

1. Are capable of understanding and have voluntarily signed the informed consent document
2. Currently receiving a stable Trogarzo-containing antiretroviral (ARV) regimen for a minimum of 3 months, and no change in background ARVs anticipated over the period of study participation; a stable regimen is defined as having no changes in dose or frequency and no interruptions greater than or equal to 2 weeks during the 3 month period
3. Have no acquired immunodeficiency syndrome (AIDS)-defining events in the 3 months before Screening, other than cutaneous Kaposi's sarcoma or wasting syndrome due to HIV
4. Are able and willing to comply with all protocol requirements and procedures
5. Are 18 years of age or older
6. Have a life expectancy that is >6 months.
7. Have a viral load <1,000 copies/mL at Screening
8. CD4+ T-cell count > 50 cells/mm3 at Screening
9. Prothrombin time (PT) and partial thromboplastin time (PTT) <1.5 times the upper limit of normal (IM Group only)

Inclusion Criteria - Healthy Volunteers (all groups):

1. Healthy volunteers born male and female as assessed by medical history and physical examination
2. Aged >18 and <50 years at the time of Screening
3. Ability and willingness to provide written informed consent
4. Willingness to comply with protocol schedule
5. Willingness to undergo HIV-1 testing
6. Non-reactive 4th generation point of care HIV-1 test at Screening
7. Hepatitis B Surface antigen negative
8. Hepatitis C antibody negative, or if reactive, Hepatitis C RNA undetectable in plasma
9. PT and PTT <1.5 times the upper limit of normal (IM Group only)
10. Volunteers born female of reproductive potential who are sexually active with a male sex partner must agree to use one effective method of contraception from the time of signing the consent to completion of the study and agree to pregnancy testing as per the schedule of events.

Volunteers born female with reproductive potential are defined as pre-menopausal volunteers born female who have not had a sterilization procedure (e.g., hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy). Volunteers born female are considered menopausal if they have not had a menses for at least 12 months and have a follicle-stimulating hormone (FSH) of greater than 40 IU/L or if FSH testing is not available, they have had amenorrhea for 24 consecutive months.

Exclusion Criteria - HIV-infected participants (all groups):

1. Any active AIDS-defining illness according to the Centers for Disease Control and Prevention (CDC) Revised Surveillance Case Definitions for HIV Infection 2008 (Morbidity and Mortality Weekly Report (MMWR) Vol.57/No. RR-10, Appendix A), or history of the same during the 3 months preceding Screening, with the following exceptions: cutaneous Kaposi's sarcoma and wasting syndrome due to HIV
2. Any significant diseases (other than HIV-1 infection) or clinically significant findings, including psychiatric and behavioral problems, determined from Screening, medical history, and/or physical examination that, in the investigator's opinion, would preclude the subject from participating in this study
3. Any significant acute illness within 1 week before the initial administration of study drug
4. Any active infection secondary to HIV requiring acute therapy; however, subjects that require maintenance therapy (i.e., secondary prophylaxis for opportunistic infections) will be eligible for the study
5. Any immunomodulating therapy (including interferon), systemic steroids, or systemic chemotherapy within 12 weeks before Enrollment
6. Any vaccination within 7 days before Day 1
7. Any female subject who either is pregnant, intends to become pregnant, or is currently breastfeeding
8. Any current alcohol or illicit drug use that, in the investigator's opinion, will interfere with the subject's ability to comply with the study schedule and protocol evaluations
9. Any radiation therapy during the 28 days before first administration of study medication
10. Any Grade 3 or 4 laboratory abnormality according to the Division of AIDS (DAIDS) grading scale, except for the following asymptomatic Grade 3 events:

    * triglyceride elevation
    * total cholesterol elevation
    * or Grade 3 or 4 reductions in levels of CD4+ T cells
11. History of coagulopathy that would preclude administration of IM injections (IM Group only)
12. Skin rashes or tattoos that would prevent ability to assess IM injection for injection-site reactions (IM Group only)
13. Use of high-dose aspirin, clopidogrel, prasugrel, ticagrelor, dipyridamole or other antiplatelet medication that would interfere with the ability to receive IM injections (IM Group only).

Exclusion Criteria - Healthy Volunteers (all groups):

1. Confirmed HIV-1 infection
2. At high risk of severe COVID-19 disease as defined by one of the following:

   * History of hypertension, atherosclerotic cardiovascular disease (ASCVD), coronary artery disease, diabetes mellitus
   * History of asthma or chronic pulmonary disease
   * History of renal disease and chronic renal insufficiency
   * BMI over 35
3. Any acute or chronic medical condition that in the opinion of the investigator would preclude participation
4. Chronic autoimmune disease
5. Active IV drug use
6. Excessive use of alcohol or recreational drugs that in the opinion of the investigator would preclude participation
7. Decompensated psychiatric illness
8. Need for chronic immunotherapy including systemic corticosteroids, other monoclonal antibody (MAb) therapy, or immunosuppressive drugs
9. Volunteers born female who are pregnant, lactating, or planning on becoming pregnant over the study period
10. Any of the following laboratory parameters:

    * Hemoglobin <10.0 g/dL
    * Absolute neutrophil count <1,000/mm3
    * Absolute lymphocyte count <500/mm3
    * Platelet count <100,000/mm3
    * Creatinine >1.25x upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) >1.5x ULN
    * Alanine aminotransferase (ALT) >1.5x ULN
    * Glucose (non-fasting) >160 mg/dL
    * Proteinuria: 2+ or greater
    * Hematuria: >10 red blood cells (RBCs) per high-power field
11. Previous receipt of an experimental MAb for HIV-1treatment or prevention in a research study
12. History of severe allergic reactions to drugs, vaccines, or drug infusion
13. Participation in another investigational clinical trial within the past 12 weeks or anticipated during the course of the current study
14. History of coagulopathy that would preclude administration of IM injections (IM Group only)
15. Skin rashes or tattoos that would prevent ability to assess IM injection for injection-site reactions (IM Group only)
16. Use of high-dose aspirin, clopidogrel, prasugrel, ticagrelor, dipyridamole any other antiplatelet medication that would interfere with the ability to receive IM injections (IM Group only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Markowitz, MD, Study Chair — TaiMed Biologics Inc. - Consultant
Locations (4):
- United States (4):
  - Anthony Mills MD Inc., Los Angeles, California
  - Gary Richmond MD, PA, Fort Lauderdale, Florida
  - Orlando Immunology Center, Orlando, Florida
  - North Texas Infectious Disease Consultants, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sentinel Group: Five (5) participants will receive two successive doses of 800mg ibalizumab administered in accordance with the prescribing information followed by five (5) successive 800mg doses on a schedule gradually increasing drug concentration and decreasing administration time.
  ibalizumab-uiyk: Ibalizumab-uiyk is an Immunoglobulin G4 (IgG4) monoclonal antibody targeting domain 2 of the extracellular portion of the Cluster of Differentiation 4 (CD4) protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Core Group-HIV+: HIV-infected Core Group participants will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via undiluted IV Push over 30 seconds. Healthy Volunteer Core Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. T
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Core Group-HIV Uninfected: Healthy Volunteer Core Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via undiluted IV Push over 30 seconds.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Intramuscular Injection Group-HIV+: HIV-infected Intramuscular Injection Group participants will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via Intramuscular Injection. Healthy Volunteer Intramuscular Injection Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via intramuscular injection.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Intramuscular Injection Group- HIV Uninfected: HIV-uninfected Intramuscular Injection Group participants will receive 2000 mg of Trogarzo followed by four (4) successive 800mg doses via IV infusion to establish a steady state which will then be followed by four doses of 800 mg of Trogarzo given by IM injection every 2 weeks.
Period: Overall Study
Arm/Group | Sentinel Group | Core Group-HIV+ | Core Group-HIV Uninfected | Intramuscular Injection Group-HIV+ | Intramuscular Injection Group- HIV Uninfected
Started | 5 | 4 | 13 | 7 | 14
Completed | 5 | 4 | 10 | 6 | 13
Not Completed | 0 | 0 | 3 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1
Not completed — non adherence to study | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sentinel Group: Five (5) participants will receive two successive doses of 800mg ibalizumab administered in accordance with the prescribing information followed by five (5) successive 800mg doses on a schedule gradually increasing drug concentration and decreasing administration time.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Core Group-HIV+: HIV-infected Core Group participants will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via undiluted IV Push over 30 seconds. Healthy Volunteer Core Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via undiluted IV Push over 30 seconds.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Core Group-HIV-uninfected: Healthy Volunteer Core Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via undiluted IV Push over 30 seconds.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Intramuscular Injection Group-uninfected: Healthy Volunteer Core Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via IM injection.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Total: Total of all reporting groups
Arm/Group | Sentinel Group | Core Group-HIV+ | Core Group-HIV-uninfected | Intramuscular Injection Group-HIV+ | Intramuscular Injection Group-uninfected | Total
Number analyzed (Participants) | 5 | 4 | 13 | 7 | 14 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (6) | 58 (6) | 31 (7) | 59 (6) | 35 (6) | 43 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 4 | 0 | 6 | 10
  Male | 5 | 4 | 9 | 7 | 8 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 8 | 2 | 6 | 18
  Not Hispanic or Latino | 5 | 2 | 5 | 4 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 2 | 4
  White | 4 | 4 | 13 | 6 | 11 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 13 | 7 | 14 | 43

OUTCOME MEASURES:

1. Primary Outcome: Safety of Trogarzo Given as IV Push Over 30 Seconds
Description: Number of subjects who complete 100% of all Trogarzo administrations given as infusion/bolus/push as per protocol
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Core Group-HIV+: HIV infected individuals will receive four (4) successive 800mg doses via undiluted IV Push over 30 seconds.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
Arm/Group | Sentinel Group | Core Group-HIV+ | Core Group-HIV Uninfected
Number analyzed (Participants) | 5 | 4 | 13
Participants | 5 | 4 | 10

2. Primary Outcome: Pharmacokinetics Bridge for IV Push and IV Infusion (Ctrough)
Description: Ratio of proportion of subjects with trough concentration (Ctrough) ≥ the threshold of 300 ng/mL given by 15 minute infusion (IVI) versus IV push (IVP) over 30 seconds
Time Frame: Day 1 infusion versus Day 85 IV Push
Population: Intent to Treat (ITT) population (Sentinel and Core participants pooled). Each participant in both the Sentinel and Core groups received IV infusion and IV push. Since the comparison between the two routes was conducted within the same participant (intra-individual comparison), data from both groups were pooled for the pharmacokinetic (PK) bridging statistical analysis. Three Core Group HIV uninfected participants discontinued prematurely and did not have IVI or IVP data.
Measure: Count of Participants; unit: Participants
Groups:
- Sentinel Group: Sentinel Group: Five (5) participants will receive two successive doses of 800mg ibalizumab administered in accordance with the prescribing information followed by five (5) successive 800mg doses on a schedule gradually increasing drug concentration and decreasing administration time.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Core Group HIV Infected: Core Group HIV infected individuals: Core group participants received an 800 mg dose of Trogarzo in accordance with the prescribing information at Day 1 and 15, and then received four (4) successive 800mg doses via undiluted IV Push over 30 seconds.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Core Group HIV Uninfected: Core Group HIV uninfected participants received a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, HIV uninfected individuals received two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via undiluted IV Push over 30 seconds.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
Arm/Group | Sentinel Group | Core Group HIV Infected | Core Group HIV Uninfected
Number analyzed (Participants) | 5 | 4 | 10
Participants
  Participants with Ctrough ≥ 300 ng/mL (IVI) | 5 | 3 | 10
  Participants with Ctrough ≥ 300 ng/mL (IVP) | 5 | 3 | 10
Statistical Analysis 1: Comparison: Sentinel Group vs Core Group HIV Infected vs Core Group HIV Uninfected; The proportion of subjects with an average Ctrough ≥ 300 ng/mL is compared between the 30-second IV push and the 15-minute IV infusion; Test type: Equivalence — The equivalence limits for the 90% confidence interval are 0.80 to 1.25. If the 90% CIs were within the equivalence limits (0.8, 1.25), it demonstrated a PK bridge between the two routes of administration; p = 1.0, Fisher Exact — H0: P1 is not different from P2; Risk Ratio (RR) = 1, 90% CI 2-sided [0.8299 to 1.2049]

3. Primary Outcome: Pharmacokinetics Bridge for IV Push and IV Infusion (AUC)
Description: Ratio of Area Under the Curve of Serum levels of Trogarzo given by 15 minute infusion versus Area Under the Curve of Serum levels of Trogarzo given by IV Push over 30 seconds
Time Frame: Day 1 infusion versus Day 85 IV Push
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Sentinel Group | Core Group HIV Infected | Core Group HIV Uninfected
Number analyzed (Participants) | 5 | 4 | 10
day*mcg/mL
  AUC (IVI) | 1232.86 (442.32) | 1143.51 (629.16) | 2772.35 (983.45)
  AUC (IVP) | 1172.95 (442.73) | 1207.62 (515.46) | 2812.55 (863.39)
Statistical Analysis 1: Comparison: Sentinel Group vs Core Group HIV Infected vs Core Group HIV Uninfected; The log transform of the ratio of the geometric means of the Area Under the Curve (AUC) for 30 second IV Push and 15 minute IV infusion is compared; Test type: Equivalence — The equivalence limits for the 90% confidence interval (CI) are 0.80 to 1.25. If the 90% CIs were within the equivalence limits (0.8, 1.25), it demonstrated a PK bridge between the two routes of administration; p = 0.5389, SAS PROC MIXED; mean geometric ratio = 1.0315, 90% CI 2-sided [0.9478 to 1.1226]

4. Primary Outcome: Safety of Trogarzo Given as an Intramuscular Injection in the Intramuscular Injection Group
Description: Number of subjects in Intramuscular Injection Group who complete 100% of all Trogarzo administrations given as infusion/bolus/push as per protocol
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Intramuscular Injection Group-HIV+: HIV-infected Intramuscular Injection Group participants will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via Intramuscular Injection.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Intramuscular Injection Group- HIV Uninfected: HIV-uninfected Intramuscular Injection Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via intramuscular injection.
Arm/Group | Intramuscular Injection Group-HIV+ | Intramuscular Injection Group- HIV Uninfected
Number analyzed (Participants) | 7 | 14
Participants | 6 | 13

5. Primary Outcome: Pharmacokinetics Bridge Demonstrated for Intramuscular Injection of Trogarzo and IV Infusion
Description: Ratio of proportion of subjects with trough concentration (Ctrough) ≥ the threshold of 300 ng/mL given by 15 minute infusion (IVI) versus intramuscular (IM) injection
Time Frame: Day 1 infusion versus Day 71 intramuscular injection
Population: ITT population (HIV+ and HIV- participants pooled). Each HIV+ and HIV- participant received IV infusion and IM. Since the comparison between the two routes was conducted within the same participant (intra-individual comparison), data from both groups were pooled for the PK bridging statistical analysis. One HIV+ participant received only the IV infusion and discontinued prematurely without receiving the IM injection.
Measure: Count of Participants; unit: Participants
Groups:
- Intramuscular Injection Group- HIV+: HIV+ participants in this group will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information at Day 1 and 15 followed by four (4) successive 800mg doses via intramuscular injection through Day 71.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Intramuscular Injection Group- HIV Uninfected: HIV- participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via intramuscular injection.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
Arm/Group | Intramuscular Injection Group- HIV+ | Intramuscular Injection Group- HIV Uninfected
Number analyzed (Participants) | 6 | 14
Participants
  Participants with Ctrough ≥ 300 ng/mL (IVI) | 5 | 14
  Participants with Ctrough ≥ 300 ng/mL (IM): number analyzed (Participants) | 6 | 13
  Participants with Ctrough ≥ 300 ng/mL (IM) | 4 | 12
Statistical Analysis 1: Comparison: Intramuscular Injection Group- HIV+ vs Intramuscular Injection Group- HIV Uninfected; The proportion of subjects with an average Ctrough ≥ 300 ng/mL is compared between IM and IV infusion; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; p = 0.34, Fisher Exact; Risk Ratio (RR) = 0.89, 90% CI 2-sided [0.69 to 1.08]

ADVERSE EVENTS:
Time Frame: Adverse events were elicited from the time of signing the informed consent through completion of the study at either day 85 (HIV+ IVP, HIV+IM, HIV uninfected IVP) or day 99 (Sentinel IVP and Uninfected IM). For HIV-uninfected individuals study duration requited establishment of an ibalizumab steady state which added 55 days to period of time over which adverse event data were collected.
Description: Adverse events were collected by subject interview, observation pre, during, and post ibalizumab infusion over 15 minute; pre, during and post ibalizumab dosing by intravenous push and pre- during, and post IM administration of ibalizumab.
Groups:
- Sentinel Group-HIV +: Five (5) participants will receive two successive doses of 800mg ibalizumab administered in accordance with the prescribing information followed by five (5) successive 800mg doses on a schedule gradually increasing drug concentration and decreasing administration time.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Core Group- HIV+: HIV-infected Core Group participants will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via undiluted IV Push over 30 seconds.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Intramuscular Injection Group-HIV+: HIV+ participants in this group will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via intramuscular injection.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
- Intramuscular Injection Group-HIV Uninfected: Healthy Volunteer Intramuscular Injection Group participants will receive a single 2000mg loading dose followed by three successive doses of 800mg in accordance with the prescribing information in order to reach steady state. Thereafter, Healthy Volunteers will receive two successive doses of 800mg ibalizumab (Trogarzo) administered in accordance with the prescribing information followed by four (4) successive 800mg doses via intramuscular injection.
  ibalizumab-uiyk: Ibalizumab-uiyk is an IgG4 monoclonal antibody targeting domain 2 of the extracellular portion of the CD4 protein. Ibalizumab-uiyk is FDA approved for the treatment of multi-drug resistant HIV in treatment experienced patients.
Arm/Group | Sentinel Group-HIV + | Core Group- HIV+ | Core Group-HIV Uninfected | Intramuscular Injection Group-HIV+ | Intramuscular Injection Group-HIV Uninfected
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/13 | 0/7 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/13 | 0/7 | 0/14
Other Adverse Events (participants affected / at risk) | 1/5 | 1/4 | 8/13 | 4/7 | 10/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentinel Group-HIV + (N=5) | Core Group- HIV+ (N=4) | Core Group-HIV Uninfected (N=13) | Intramuscular Injection Group-HIV+ (N=7) | Intramuscular Injection Group-HIV Uninfected (N=14)
otitis media (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (7)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
allergic rhinitis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
injection site pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hyperglycemia (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hematoma at infusion site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
bruising (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Limitations of the trial include::

1. difficulty in recruitment of HIV-infected individuals who were using ibalizumab as part of a suppressive regimen as issues with continued supply and reimbursement emerged necessitating the recruitment of HIV-uninfected participants in whom the pharmacokinetics of ibalizumab differ from the HIV-infected population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data are considered the property of the sponsor and cannot be published without sponsor authorization. The sponsor agrees to work with the PI to determine how any manuscript is written and edited and the publication to which it is submitted. The sponsor has the authority of final determination in these matters.

DOCUMENTS (2):
  • Study Protocol (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT03913195/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT03913195/SAP_002.pdf